CLINICAL TRIAL: NCT03140358
Title: The Use of Atropine 0.01% in the Prevention and Control of Myopia (ATOM3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Audrey Chia Wei-Lin, Adjuct Associate Professor, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1359/45/2016
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Premyopia atropine (Active Comparator): On Atropine 0.01%
  Interventions: Drug: Atropine sulfate 0.01%
- Premyopia placebo (Placebo Comparator): On placebo
  Interventions: Drug: Placebo
- Low myopia atropine (Active Comparator): On Atropine 0.01% daily or every other day
  Interventions: Drug: Atropine sulfate 0.01%
- Low myopia placebo (Placebo Comparator): On placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine sulfate 0.01% — Atropine 0.01%
  Arms: Low myopia atropine; Premyopia atropine
Drug: Placebo — placebo
  Arms: Low myopia placebo; Premyopia placebo

SUMMARY:
Study of low dose atropine in preventing the onset and progression of myopia in high risk children with pre-myopia or low-myopia.

DETAILED DESCRIPTION:
High risk children (with family history of myopia) with low hyperopia or low myopia will be randomized to atropine or placebo, with 2 -2.5 year treatment and 1 year washout.

ELIGIBILITY:
Inclusion criteria

1. One parent with myopia (<-3D in at least one eye)
2. SE +1.00D to -1.50D
3. Astigmatism < = 1.50D
4. Distance vision logMAR 0.2 or better in both eyes
5. Intraocular pressure of not greater than 21 mmHg
6. No allergy to atropine, cyclopentolate, proparacaine and benzalkonium chloride

Exclusion Criteria:

1. Any eye or systemic disease that affect vision or refractive error
2. Conditions where topical atropine contraindicated
3. Previous use of atropine or pirenzepine
4. Known past/current amblyopia or strabismus

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Spherical Equivalent | 3.5 years
  SE

SECONDARY OUTCOMES:
Axial Length | 3.5 years
  AL

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Chia, Principal Investigator — Singapore National Eye Center
Locations (1):
- Singapore eye research institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No